CLINICAL TRIAL: NCT04995354
Title: Self Healing Gel as a Vehicle for Recombinant Human Epidermal Growth Factor in Treatment of Oral Mucositis Following Cancer Therapy
Brief Title: Efficacy of EGF-loaded Self Healing Gel in Treatment of Oral Mucositis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Basma Elsaadany, Lecturer of oral medicine and periodontology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MucoCU
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis | interventions — Hydrogels

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Containers supplied for groups I and II will be identical and will be supplied by a third party pharmacist not a member of this study to ensure participant and patient blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EGF loaded Hydrogel (Gp I) (Experimental): 30 patients will receive EGF loaded Hydrogel (Intervention 1) to be applied three times a day for 1weeks.
  Interventions: Drug: EGF loaded Hydrogel
- Hydrogel alone ( Gp II) (Active Comparator): 30 patients will receive Hydrogel alone (Intervention 2) to be applied three times a day for 2 weeks.
  Interventions: Drug: Hydrogel
- Control (Gp III) (No Intervention): 30 patients will receive the standard of care treatment (Control) which includes benzydamine mouthwash, increased hydration, topical analgesics and antifungals.

INTERVENTIONS:
Drug: EGF loaded Hydrogel — Patients will receive 25 Ug/day of EGF. This is the estimated daily dose that will be obtained when the patient applies the gel thrice daily. Patients will receive the treatment for one week
  Other Names: Epidermal Growth Factor-loaded Hydrogel
  Arms: EGF loaded Hydrogel (Gp I)
Drug: Hydrogel — Non-medicated self-healing hydrogel to be applied three times a day for 1 week
  Other Names: Self-healing Hydrogel
  Arms: Hydrogel alone ( Gp II)

SUMMARY:
Cancer treatment, including radiation along with aggressive chemotherapy, increases the patient's survival rate. However, they possess toxic side effects. Oral mucositis is one of the most serious complications of cancer treatment, which occurs in most of patients receiving cancer therapy. Mucositis can dramatically affect the patient's quality of life .Epidermal growth factor (EGF) is a dominant factor in early keratinocyte differentiation, proliferation and migration. However, a major obstacle in most studies is that there isn't prolonged contact between the applied treatment and the oral mucosa to achieve the optimum therapeutic effect. Thus, a new vehicle for EGF is needed to achieve sufficient prolonged contact with oral mucosa. The present project aims at employing EGF as therapeutic agent for mucositis dealing with the challenges of delivery of such macromolecule to the oral mucosa by using self-healing gels to maximize the drug effect.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are those over 18 years of age with WHO grade 3 or 4 oral mucositis receiving radio- or chemotherapy as treatment for head and neck cancer.

Exclusion Criteria:

* Patients with hematologic malignancies or those with known allergic reactions to the drug.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
The European Organization for Research and Treatment of Cancer Quality of Life questionnaire | Baseline
  Questionnaire developed to assess the quality of life of cancer patients. The questionnaire used will be for that for head and neck patients (EORTC QLQ - H&N43) https://www.eortc.org/app/uploads/sites/2/2018/08/Specimen-HN43-English.pdf
WHO grade of mucositis | Baseline
  Grade 1 Soreness, with or without erythema
  Grade 2 Erythema, ulcers; still able to swallow solid foods
  Grade 3 Ulcers with extensive erythema; unable to swallow solid foods
  Grade 4 Ulcers with extensive erythema; alimentation not possible
The European Organization for Research and Treatment of Cancer Quality of Life questionnaire | After 7 days of treatment
  Questionnaire developed to assess the quality of life of cancer patients. The questionnaire used will be for that for head and neck patients (EORTC QLQ - H&N43) https://www.eortc.org/app/uploads/sites/2/2018/08/Specimen-HN43-English.pdf
WHO grade of mucositis | After 7 days of treatment
  Grade 1 Soreness, with or without erythema
  Grade 2 Erythema, ulcers; still able to swallow solid foods
  Grade 3 Ulcers with extensive erythema; unable to swallow solid foods
  Grade 4 Ulcers with extensive erythema; alimentation not possible
The European Organization for Research and Treatment of Cancer Quality of Life questionnaire | After 14 days of treatment.
  Questionnaire developed to assess the quality of life of cancer patients. The questionnaire used will be for that for head and neck patients (EORTC QLQ - H&N43) https://www.eortc.org/app/uploads/sites/2/2018/08/Specimen-HN43-English.pdf
WHO grade of mucositis | After 14 days of treatment.
  Grade 1 Soreness, with or without erythema
  Grade 2 Erythema, ulcers; still able to swallow solid foods
  Grade 3 Ulcers with extensive erythema; unable to swallow solid foods
  Grade 4 Ulcers with extensive erythema; alimentation not possible

CONTACTS AND LOCATIONS:
Overall Officials: Basma AA Zakaria, PhD, Principal Investigator — Lecturer at the Faculty of Dentistry - Cairo University

IPD SHARING:
Plan to Share IPD: No